CLINICAL TRIAL: NCT00283582
Title: Randomized Double-blind Placebo-controlled Trial of Primary Prophylaxis With Recombinant Human Thrombopoietin Administered to Patients With High Risk Sarcoma Receiving Intensive Chemotherapy
Brief Title: Trial of Primary Prophylaxis With rhTPO Administered to Patients With High Risk Sarcoma Receiving Intensive Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: DM00-435
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

INTERVENTIONS:
Drug: rhTPO

SUMMARY:
Intensive chemotherapy is often associated with low platelet counts often requiring platelet transfusions to maintain platelet counts. In previous clinical studies administration of rhTPO has been demonstrated to increase platelet counts.

DETAILED DESCRIPTION:
To evaluate the effectiveness of intravenous rhTPO vs. placebo as primary prophylaxis in reducing the cumulative proportion of patients requiring platelet transfusion for severe chemotherapy-induced thrombocytopenia (platelet count <15,000) during the first four study cycles. To evaluate the severity and duration of thrombocytopenia and neutropenia associated with rhTPO prophylaxis, the impact of rhTPO prophylaxis on health economics/cost effectiveness, and patient quality of life. To assess the safety of multiple IV doses of rhTPO.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed new diagnosis of moderate or high-grade sarcoma (except leiomyosarcoma of gastrointestinal origin)
* Must have high risk disease by American Joint Committee on Cancer (AJCC) Staging System Stage IIC, III, or IV
* Must have recovered from surgery for a minimum of 2 weeks
* Must be scheduled for a minimum of 4 cycles of AI therapy
* Must be 13 years or older
* Must have ECOG performance status of 0, 1, or 2.
* Must have life expectancy of at least 12 weeks.
* Left ventricular ejection fraction must be more than 50%.
* Laboratory data within normal limits.

Exclusion Criteria:

* Prior front-line standard or experimental therapy for sarcoma
* History of bone marrow and or peripheral blood progenitor cell transplantation
* Prior pelvic radiation or radiation therapy to more than 25% of bone marrow reserves
* Prior treatment with megakaryocyte growth and differentiation factor
* Prior treatment with rhTPO
* History of platelet disorder
* History of myocardial infarction, stroke, pulmonary embolism, or deep vein thrombosis within the past 12 months
* Pregnant or lactating women
* Use of anticoagulants such as coumadin, heparin, etc.
* Known HIV or hepatitis

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
CBC with diff. at least three times a week and daily if platelet less than 50,000. Chemistry, coagulation, urinalysis performed at baseline and at end of cycle if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, M.D., Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org